CLINICAL TRIAL: NCT01520103
Title: Randomized Phase II Study to Compare Vinorelbine In Combination With the mTOR Inhibitor Everolimus vs. Vinorelbin Monotherapy for Second-line Treatment in Advanced Breast Cancer
Brief Title: Study to Compare Vinorelbine In Combination With the mTOR Inhibitor Everolimus vs. Vinorelbin Monotherapy for Second-line Treatment in Advanced Breast Cancer
Acronym: VicTORia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: iOMEDICO AG (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-MAM-0110; 2011-001024-38 (EudraCT Number); CRAD001JDE38T (Other: Novartis Pharma GmbH)
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Her2-negative Metastatic Breast Cancer; Her2-negative Locally Advanced Breast Cancer
Keywords: Metastatic breast cancer; locally advanced breast cancer; Her2/new negative; HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vinorelbin and Everolimus (Experimental)
  Interventions: Drug: Vinorebine, Everolimus
- standard therapy (Other): Vinorelbin
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorebine, Everolimus — Vinorelbin: i.v. 25 mg/ m² d1, d8, d15 3qw Everolimus: oral 5 mg/d d1-21 3qw until progress
  Arms: Vinorelbin and Everolimus
Drug: Vinorelbine — Vinorelbin: i.v. 25 mg/ m² d1, d8, d15 3qw until progress
  Arms: standard therapy

SUMMARY:
The purpose of this study is Examination of the superiority of a combination of vinorelbine with the mTOR Inhibitor Everolimus vs. vinorelbine monotherapy for second-line treatment in advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1 .Dated and signed patient informed consent before start of any in the protocol specified procedures 2. Histologically or cytologically confirmed Her2/neu negative, metastatic or locally advanced breast cancer, including inoperable local relapse, with measurable or non-measurable lesions for which

* a palliative second line chemotherapy is indicated. Antihormone palliative pretreatments do not count as separate treatment lines
* treatment with anthracycline and/or taxanes has failed or is not suitable
* which cannot be adequately treated by operation or radiotherapy on its own 3. An exclusive anti-hormone therapy is not indicated for the patient 4. ECOG Performance Status of 0-2 5. Women >= 18 years of age 6. Life expectancy of at least 12 weeks 7. Adequate bone marrow, liver and renal function (according to SmPC of Vinorelbine, Afinitor®) based on laboratory assessments raised within 7 days prior to start of study treatment:
* Haemoglobin >= 9.0 g/dl
* Absolute neutrophil count (ANC) >= 2/mm³
* Thrombocytes >= 100/µl
* INR >= 2
* Serum bilirubin =< 1.5x upper limit of normal ( in patients with known Gilbert syndrome, total bilirubin =< 3x upper limit of normal, with direct bilirubin =< 1.5x upper limit of normal
* ALT and AST =< 2.5x upper limit of normal (=< 5x upper limit of normal in subjects with liver metastases)
* Serum cholesterol =< 300 mg/dl or 7.75 mmol/l and triglycerides =< 2.5x upper limit of normal (with lipid lowering drugs permitted)
* Serum creatinin =< 2x upper limit of normal 8. Documentation of a negative pregnancy test in women of childbearing potential within 7 days prior to start of study. Sexual active pre-menopausal women are required to use adequate contraception throughout the duration of the study, except for oestrogen containing contraceptives

Exclusion Criteria:

1. Previous treatment with Vinorelbine or an inhibitor of mTOR
2. Treatment with other study medication within 28 days before start of treatment
3. Patients who have received prior radiotherapy to ≥ 25% of the bone marrow
4. Other tumours in the previous 5 years with exception of an adequately treated basal cell carcinoma of the skin or a preinvasive cervix carcinoma
5. Simultaneous use of known CYP3A4 inducers (e.g. Phenytoin, Rifampicin) or inhibitors of this enzyme (e.g. Itraconazole, Ketoconazole), therefore also use of mistletoe, St John's wort or grapefruit juice
6. Patients to whom at least one of the conditions applies:

   * Substance abuse
   * medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
   * Legal incapacity or limited legal capacity
   * Subjects who are unable to take oral medication
   * Any condition that could jeopardise the safety of the patient and their compliance in the study as judged by the investigator
7. History of cardiac dysfunction including one of the following:

   * Myocardial infarction by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function
   * History of documented congestive heart failure (NYHA ≥ 3)
   * Documented cardiomyopathy
8. Known HIV infection or chronic hepatitis B or C or history of hepatitis B / C
9. Active clinically relevant infection (> grade 2 NCI-CTC Version 4.03)
10. Clinical or radiological detection of CNS metastases
11. Patients receiving concomitant immunosuppressive agents or chronic use of corticosteroids at the time of study entry except in cases outlined below:

    * topical applications (e.g. rash,) inhaled sprays, (e.g. obstructive airway diseases) eye drops or local injections (e.g. intraarticular) are allowed
12. Active bleeding diathesis or an oral anti-vitamin K medication (except low-dose warfarin and aspirin or equivalent, as long as the INR ≤ 2)
13. Kidney function disorder requiring dialysis
14. Seriously impaired liver function (Child-Pugh, class C)
15. Known hypersensitivity reaction to Vinorelbine or Everolimus
16. Pregnant or breast-feeding subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Assessment over 36 months, minimum 12 month
  Progression-free survival (PFS) will be defined as the time from randomization to the time of disease progression or relapse or death.

SECONDARY OUTCOMES:
Safety and tolerability | Assessment over 36 months
  Capture all adverse events, serious adverse events, all side effects of the study medication, serious side effects, adverse events that lead to temporary or complete discontinuation of the study treatment and the Rates and causes of death.
  A safety interims analysis is planned, as soon as 60 subjects have finished at least two treatment cycles.
Rate of Progression Free Survival after 6 months (6 months PFSR) | Assessment over 36 months
  descriptive Evaluation, for the monotherapy (arm 2) a median PFS of 4 months is assumed. It is expected that the combination therapy will prolong the median PFS to 6.5 months.
Overall survival (OS) | 36 months
  The duration of overall survival (OS) will be determined by measuring the time interval from randomization to the date of death or last observation.
Response rate (CR, PR) | 36 months
  The tumour status of patients will be evaluated nine weekly during the treatment until detection of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lerchenmüller, Dr., Principal Investigator — Hämatologisch-onkologische Gemeinschaftspraxis, Münster
Locations (1):
- Hämatologisch-onkologische Gemeinschaftspraxis, Münster, Münster, Germany

REFERENCES:
- [Derived] Decker T, Marschner N, Muendlein A, Welt A, Hagen V, Rauh J, Schroder H, Jaehnig P, Potthoff K, Lerchenmuller C. VicTORia: a randomised phase II study to compare vinorelbine in combination with the mTOR inhibitor everolimus versus vinorelbine monotherapy for second-line chemotherapy in advanced HER2-negative breast cancer. Breast Cancer Res Treat. 2019 Aug;176(3):637-647. doi: 10.1007/s10549-019-05280-2. Epub 2019 May 21. PMID 31115844
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de